CLINICAL TRIAL: NCT04424472
Title: Assessing the Utility of Ultrasound Compared to Cross-Sectional Imaging in the Follow-up of Patients With Renal Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00145327
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ultrasonography

STUDY DESIGN:
Masking Description: The sonographer for the additional ultrasound will be blinded as will be the blinded radiology who will compare the US to the most recent negative CT/MRI to determine if recurrence is visualized by US
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasonography (Experimental): Patient will be scheduled to undergo an additional US by a blinded sonographer within 4 weeks of their most recent cross-sectional imaging that indicated a recurrence
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Abdominal Ultrasonography

SUMMARY:
The aim of this study is to determine the utility of renal ultrasonography (US) in the detection of abdominal recurrences after definitive therapy for renal cell carcinoma (RCC) and compare the detection rate to that of cross-sectional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 year of age or older.
* Patients having undergone radical or partial nephrectomy for the indication of renal cell carcinoma.
* Most recent imaging study must have been either computed tomography (CT) or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Patients with pT4 disease (tumor invades beyond the Gerota fascia: including contiguous extension into the ipsilateral adrenal gland).
* Patients with metastatic disease prior to time of surgery requiring systemic treatment.
* Patients with another active cancer diagnosis requiring systemic treatment.
* Patients with contrast allergies.
* Patients with baseline chronic kidney disease (GFR < 45 ml/min/1.73 m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Utility of Renal Ultrasonography (US) in the detection of abdominal recurrences | 4 weeks
  Renal Cell Carcinoma (RCC) recurrence detection of ultrasonography in patients who have undergo definitive therapy for RCC compared to detection rate of cross-sectional imaging

SECONDARY OUTCOMES:
Radiation Burden | 5 years
  Compare the average radiation exposure over 5 years for patients on current standard of care imaging surveillance for RCC, which consists of both ultrasound and cross-sectional imaging, to that of patients who would only receive cross-section imaging surveillance for RCC. This would yield overall increase in radiation burden for patients with RCC

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No